CLINICAL TRIAL: NCT03333954
Title: Feasibility Study of Compensation for Blindness With the PRIMA System in Patients With Dry Age Related Macular Degeneration
Acronym: PRIMA FS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Science Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-PRIMA-FS
Record Dates: First submitted 2017-10-27; First posted 2017-11-07 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-02

CONDITIONS: Dry Age-related Macular Degeneration
Keywords: atrophic macular degeneration; geographic atrophy; macular degeneration; dry macular degeneration; AMD; retina implant; retinal prosthesis; visual prosthesis
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: PRIMA — The PRIMA Bionic Vision System is a device for treatment of patients who have lost their sight through outer retinal degenerative conditions of the eye such as atrophic dry age related macular degeneration.
  The PRIMA System is designed to provide partial restoration of the patient's visual function through electrical stimulation of the retinal neurons by a sub-retinally implanted stimulator that replace part of the degenerate photoreceptors

SUMMARY:
In this study, the principle functionality of the device will be tested in humans for the first time. The study will evaluate the extent to which patients with atrophic dry age related macular degeneration (AMD) have evoked light perception using the implant.

DETAILED DESCRIPTION:
In this study subjects are provided with a PRIMA sub-retinal implant in one eye. A camera integrated in the external components of the implant captures visual information of the environment, this information is processed by a pocket processor and then transmitted via projected IR light onto the implant. The implant received the projected IR light and stimulates the nerve cells of the retina. Interim analysis will be performed at 6 months after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Is 60 years or older at the date of enrolment;
* Has a confirmed diagnosis of advanced dry age related macular degeneration with an atrophy size of at least 3 optic disc diameters;
* Has best corrected visual acuity of the study eye of logMAR 1.3 (20/400) or worse measured by ETDRS;
* Has no foveal perception measured by micro-perimetry in the study eye (≤ 4 dB on Opko scale or equivalent) ;
* Has a study eye that is able to perceive light;
* Has useful vision on the non-study eye;
* Has a refraction of study eye between -3 and + 4 (limits included) for patient with IOL (there is no refraction criteria for patients with natural lens);
* Understands and accepts the obligation to present for all schedule follow-up visits.
* Patient signed informed consent

Exclusion Criteria:

* Has cataracts that may influence the visual function of the study eye;
* Has an aphakic study eye
* Had cataract surgery in the last 1 month;
* Active sub-macular choroidal neovascularization in the study eye;
* Has any disease (other than study allowed diseases) or condition that affects retinal function of the study eye (e.g., central retinal artery/vein occlusion, end-stage diabetic retinopathy, retinal detachment, infectious or inflammatory retinal disease, severe glaucoma, optic neuropathy, myopic chorio-retinal atrophy etc.);
* Has an implanted telescope in one eye;
* Has any disease or condition that prevents adequate examination of the study eye including, but not limited to, corneal degeneration that cannot be resolved prior to implantation. Note, that this criterion is also important for the function of the implant;
* Has an endothelia cell count of less than 1000 cells/mm² in the study eye;
* Suffers from nystagmus;
* Has any disease or condition that precludes the understanding or communication of the informed consent, study requirements or test protocols (e.g., deafness, severe multiple sclerosis, amyotrophic lateral sclerosis, severe neuritis, etc);
* Has a history of epileptic seizure;
* Has a history of chronic or recurrent infection or inflammation that would preclude participation in the study;
* Has a known sensitivity to the contact materials of the implant (iridium oxide, silicon-carbide and titanium);
* Presents with hypotony in the study eye;
* Presents with hypertony in the study eye;
* Has another active implanted device (e.g. cochlear implant, pacemaker) that may interfere with the device function, or diagnoses requiring such an active implant;
* Has active cancer or a history of intraocular, optic nerve or brain cancer and metastasis;
* Is an immune-suppressed subject (e.g., due to HIV positive diagnosis, etc.);
* Is carrier of multi-resistant germs;
* Is receiving anticoagulation therapy that cannot be adapted to allow eye surgery;
* Is participating in another investigational drug or device study that may interfere with the present study;
* Patients with recurrent or chronic inflammations or infections are excluded from the study. Specifically, patients with the following disorders are excluded:

  * Common inflammation - severe chronic and consuming diseases that frequently associated with infection (e.g. Crohn disease, Whipple's disease);
  * Active inflammation in the area of the eye (e.g. herpes of cornea and/or conjunctiva, recurrent blepharoconjunctivitis, hordeolum, chalazion);
* Has a severe psychological disorder. When in any doubt, an expert assessment needs to be arranged to clarify whether the patient's psychological health is suitable for the trial. In any doubts of the subjects psychological status a clinical psychologist, psychologist or the community doctor/general practitioner should be involved. The patient must have the legal capacity to sign the informed consent;
* Has severe renal, cardiac, hepatic etc. organ diseases;
* Has head dimension that are incompatible with the Visual Interface.
* Has too high and unrealistic expectation (e.g., believes that a benefit is guaranteed or expect normal vision after surgery)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Elicitation of perception | 6 months after implantation
  Elicitation of visual perception by electrical stimulation of the PRIMA implant measured by Octopus Visual Field
Elicitation of perception | 6 weeks after implantation
  Elicitation of visual perception by electrical stimulation of the PRIMA implant measured by Octopus Visual Field
Elicitation of perception | 3 months after implantation
  Elicitation of visual perception by electrical stimulation of the PRIMA implant measured by Octopus Visual Field
Elicitation of perception | 12 months after implantation
  Elicitation of visual perception by electrical stimulation of the PRIMA implant measured by Octopus Visual Field
Elicitation of perception | 18 months after implantation
  Elicitation of visual perception by electrical stimulation of the PRIMA implant measured by Octopus Visual Field
Elicitation of perception | 24 months after implantation
  Elicitation of visual perception by electrical stimulation of the PRIMA implant measured by Octopus Visual Field
Elicitation of perception | 36 months after implantation
  Elicitation of visual perception by electrical stimulation of the PRIMA implant measured by Octopus Visual Field

SECONDARY OUTCOMES:
Visual Acuity | 18, 24 and 36 months after implantation if applicable
  Visual acuity is a measure of the ability of the visual system to distinguish shapes and details of objects at a given distance. This study use the Landolt Ring to measure visual acuity
Letter Visual Acuity | 48, 60 and 72 month after implantation
  Visual acuity is a measure of the ability of the visual system to distinguish shapes and details of objects at a given distance. This endpoint use the ETDRS charts to measure visual acuity
Quality of Live measured by IVI | 48, 60 and 72 month after implantation
  IVI-Impact of Vision Impairment questionnaire (quality of life based on patient reported outcome of functional vision, participation in vision-related daily living activities and emotional well-being)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A. De Rothschild/ Hopital des Quinze Vingts/, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muqit MMK, Le Mer Y, Olmos de Koo L, Holz FG, Sahel JA, Palanker D. Prosthetic Visual Acuity with the PRIMA Subretinal Microchip in Patients with Atrophic Age-Related Macular Degeneration at 4 Years Follow-up. Ophthalmol Sci. 2024 Mar 7;4(5):100510. doi: 10.1016/j.xops.2024.100510. eCollection 2024 Sep-Oct. PMID 38881600
- [Derived] Muqit M, Mer YL, de Koo LO, Holz FG, Sahel JA, Palanker D. Prosthetic Visual Acuity with the PRIMA System in Patients with Atrophic Age-related Macular Degeneration at 4 years follow-up. medRxiv [Preprint]. 2023 Nov 13:2023.11.12.23298227. doi: 10.1101/2023.11.12.23298227. PMID 38014146
- [Derived] Palanker D, Le Mer Y, Mohand-Said S, Sahel JA. Simultaneous perception of prosthetic and natural vision in AMD patients. Nat Commun. 2022 Jan 26;13(1):513. doi: 10.1038/s41467-022-28125-x. PMID 35082313
- [Derived] Palanker D, Le Mer Y, Mohand-Said S, Muqit M, Sahel JA. Photovoltaic Restoration of Central Vision in Atrophic Age-Related Macular Degeneration. Ophthalmology. 2020 Aug;127(8):1097-1104. doi: 10.1016/j.ophtha.2020.02.024. Epub 2020 Feb 25. PMID 32249038